CLINICAL TRIAL: NCT00504036
Title: Medico Economic Evaluation of a Temporary (6 Months) Intra-gastric Balloon in Morbidly Obese Patients Before a Gastric By-pass. A Randomised Multicenter Study Comparing the Usual Strategy to Two Types of Gastric Balloon
Brief Title: Efficacy of Preoperative Intra Gastric Balloon in Morbidly Obese Patients Selected for Gastric By-pass
Acronym: BIGPOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060408
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2008-10

CONDITIONS: Morbid Obesity
Keywords: Obesity; Morbid obesity; Gastric balloon; Gastric by-pass; Morbid obesity with BMI > 45 kg/m²
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-gastric balloon (Experimental): Patients will receive either an air-filled or water-filled intra-gastric balloon.
  Interventions: Device: inflatable intra-gastric balloon
- Usual care (No Intervention): Usual care will be given to the patients.

INTERVENTIONS:
Device: inflatable intra-gastric balloon — inflatable intra-gastric balloon
  Arms: Intra-gastric balloon

SUMMARY:
To demonstrate, during a prospective randomized medico-economic study, in morbidly obese patients (BMI > 45 kg/m²) selected for a laparoscopic gastric by-pass that, in comparison to usual care, a temporary intra-gastric balloon (6 months) decreases medical costs and peri-operative morbidity.

DETAILED DESCRIPTION:
On inclusion, comorbidities associated with obesity will be recorded. After recording of the informed consent patients will be randomized in two groups: usual care or intra-gastric balloon. In the latter, a second randomization will be performed between air-filled balloon or water-filled balloon. Six months later, after withdrawal of the balloon (if required), laparoscopic gastric by-pass will be performed. Thereafter, patients will be followed during 6 months.

On each visit, inclusion, 3 months, 6 months, surgery, 1 month and 6 months post surgery, a medical and biological evaluation will be systematically performed.

The main criteria of judgement is the rate of admission in ICU during more than 24 hrs during the 30 days following surgery.

The secondary criteria of judgement is: the differences in pre-operative weight loss between the 2 groups, number of complications occurring during the 30 days after surgery, differences in different scales of quality of life (SF36, IWQOL-lite), differences in operative time, length of hospital stay, readmissions, and medical cots between the two strategies. Efficacy and tolerance of each type of balloon (air-filled or water-filled) will be compared in the intra-gastric balloon group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Patients with morbid obesity with BMI > 45 kg/m² requiring a gastric by-pass by laparoscopy.
* No efficacy of previous treatment on obesity
* Firmed informed consent

Exclusion Criteria:

* Patients in whom laparoscopy is contra-indicated
* Indication of gastric by-pass by laparoscopy retained without multidisciplinary advice
* Morbid obesity present since less than 5 years
* Severe associated pathology, non-related to obesity, impairing vital prognosis on a short or mean time
* Past history of gastric surgery, or gastric complication related to gastric lap-band
* Lack of health insurance
* Patient refusing to be followed 6 months before and after surgery
* Drug abuse
* Pregnancy or foreseeable pregnancy during the study
* Patients taking anticoagulant agents or steroids
* Patients with hiatal hernia > 4 cm
* Patients with active ulcerated esophagitis (grade C-D in Los Angeles Classification)
* Patients with duodenal or gastric ulcer
* Patients with gastric or esophageal varices
* Patients with NSAIDs not taking PPI
* Patients with bulimia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Rate of admission in Intensive Care Units | > 24 hrs during the 30-day period following gastric by-pass

SECONDARY OUTCOMES:
Differences in absolute weight loss | at 6 months, before gastric by-pass, between the 2 strategies
Number and types of complications occurring | during the 30-day post-operative period
Number of comorbidities present | after the 6-month initial period
Differences in quality of life | at the end of first 6-month period and at the end of the study
Differences in time of surgery, length of stay, readmission | during the 30-day post by-pass period
Differences in medical costs between the 2 strategies | 6 months before and after gastric by-pass

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Coffin, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Louis Mourier, Colombes, France

REFERENCES:
- [Result] Fernandes M, Atallah AN, Soares BG, Humberto S, Guimaraes S, Matos D, Monteiro L, Richter B. Intragastric balloon for obesity. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD004931. doi: 10.1002/14651858.CD004931.pub2. PMID 17253531